CLINICAL TRIAL: NCT01631045
Title: The Effect of a Meal on Brain Activation in Reward Pathways
Acronym: Satiety
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Assistant Professor, University of Washington
Other Study IDs: 38022
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Brain Response to Visual Food Cues
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- 15 min: Subjects post-meal brain MRI will be 15 minutes after breakfast.
- 30 min: Subjects post-meal brain MRI will be 30 minutes after breakfast.
- 60: Subjects post-meal brain MRI will be 60 minutes after breakfast.
- 120: Subjects post-meal brain MRI will be 120 minutes after breakfast.
- 180: Subjects post-meal brain MRI will be 180 minutes after breakfast.
- 240: Subjects post-meal brain MRI will be 240 minutes after breakfast.
- 300: Subjects post-meal brain MRI will be 300 minutes after breakfast.

SUMMARY:
Scientists have studied how fasting and nutrients affect brain function in animals. The purpose of this study is to look at the effects of both fasting and food intake on brain function and memory in humans. To do this the investigators will use functional MRI to observe the brain and its function while fasting and after a meal. Understanding the action of these hormones in the brain may eventually lead to new ways to help people avoid obesity or lose weight.

DETAILED DESCRIPTION:
Potential subjects will participate in a short phone screening interview and if eligible, will come to the University of Washington hospital 2 times. At the first health screening visit, we will go over the subjects' medical history, weight and height, and eating habits. This visit will take an hour or so and eligible subjects will then schedule the study visit. For the study visit, subjects will have to fast overnight from 9:30 pm the night before and arrive at the hospital at 8:00am. At 8:30 am, the subject will have a 30 minute MRI scan of the brain done in the University of Washington Radiology Department. During the MRI scan they will see pictures of common objects and foods and be asked to remember the photos they saw. At 9 am subjects will eat a standard breakfast, and they will not eat again until after the second MRI. The time of their second MRI will be randomly assigned to one of seven time points anywhere from 15 minutes to 5 hours after the breakfast. After the MRI, subjects will be allowed to eat freely from food we provide. Subjects will receive $10 for the health screening visit, and $50-85 depending on the length of the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50
2. Body mass index (BMI) 18.5-24.9 kg/m2

   * Age and weight are restricted because of known changes in appetite and satiety with aging and changes in body weight.

Exclusion Criteria:

1. Current dieting for weight loss or restrained eating
2. History of eating disorders, prior obesity, or weight loss surgery
3. Chronic health conditions, including diabetes
4. Use of medications that alter appetite (e.g., atypical anti-psychotics)
5. Pregnancy or use of oral contraceptives of estrogen replacement
6. Participation in other studies that might affect appetite or body weight
7. Recreational drug use or alcohol use of >2 drinks per day
8. Food allergies to study foods or inability to taste
9. Current smoker
10. Any contraindications to MRI such as implanted metal of claustrophobia

    * Current dieting, restrained eating, eating disorders, prior weight loss surgery, diabetes, chronic disease (e.g., cardiovascular disease, cancer), and estrogen use are restricted or excluded due to documented influences on the hormones of interest. Smokers and regular alcohol users are excluded consistent with prior studies of appetite regulation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will enroll 21 healthy subjects. Participants will be recruited by flyers posted at the University and by newspaper advertisements.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
BOLD response as measured by brain fMRI during viewing of food photographs | We will randomly assign subjects to one of 7 timepoints for a post-meal brain MRI - 15, 30, 60, 120, 180, 240, or 300 minutes after their breakfast.
  To determine whether the change in brain response (as captured by MRI) to visual food cues with food intake is a marker of satiety. We hypothesize that consumption of a meal will reduce brain activation by food cues and that these reductions will be temporally associated with both subjective and objective measures of satiety.

SECONDARY OUTCOMES:
Secondary endpoints are the amount of food eaten at a lunch buffet and self-reported appetite ratings. | Every 30 minutes throughout study.
  To measure subjective appetite and satiety, subjects will complete serial visual analog rating scales (VAS) of hunger and fullness every 30 minutes. We predict that the percentage change in brain activation will correlate with changes in self-reported hunger and fullness. After the post-meal scan, we will obtain measurements of objective satiety for each subject by monitoring his or her food intake during a 30 minute ad libitum buffet meal. The buffet will be surreptitiously monitored, allowing us to assess ad libitum caloric intake and food choices.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Schur, MD, MS, Principal Investigator — Assistant Professor
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Mehta S, Melhorn SJ, Smeraglio A, Tyagi V, Grabowski T, Schwartz MW, Schur EA. Regional brain response to visual food cues is a marker of satiety that predicts food choice. Am J Clin Nutr. 2012 Nov;96(5):989-99. doi: 10.3945/ajcn.112.042341. Epub 2012 Sep 18. PMID 22990034